CLINICAL TRIAL: NCT03760809
Title: The Effect of Different Dose of Dexmedetomidine Combined With Hydromorphone in Children With Tonsillectomy and Adenoidectomy
Brief Title: Dexmedetomidine Combined With Hydromorphone in Tonsillectomy and Adenoidectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: dex-hyd
Record Dates: First submitted 2018-11-20; First posted 2018-11-30 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2019-04

CONDITIONS: Agitated; State, Acute Reaction to Stress
Keywords: dexmedetomidine; hydromophine; tonsillectomy and adenoidectomy
MeSH Terms: conditions — Psychomotor Agitation; Stress Disorders, Traumatic, Acute | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): Dexmedetomidine(0.5 μg／kg)/hydromophine-based general anesthesia
  Interventions: Drug: Dexmedetomidine 0.5μg／kg
- group B (Experimental): Dexmedetomidine(1μg／kg)/hydromophine-based general anesthesia
  Interventions: Drug: Dexmedetomidine 1μg／kg

INTERVENTIONS:
Drug: Dexmedetomidine 0.5μg／kg — Group A received dexmedetomidine 0.5μg／kg (diluted to 100ml，influded in 5 mins at the beginning of the surgery) and hydromophine 0.03 mg／kg as a bolus.
  Other Names: Dexmedetomidine Hydrochloride Injection
  Arms: group A
Drug: Dexmedetomidine 1μg／kg — Group B received dexmedetomidine 1μg／kg (diluted to 100ml，influded in 5 mins at the beginning of the surgery) and hydromophine 0.03 mg／kg as a bolus.
  Other Names: Dexmedetomidine Hydrochloride Injection
  Arms: group B

SUMMARY:
Tonsillectomy and adenoidectomy is one of the most common pediatric surgeries, and agitation and severe postoperative pain have been considered a very common complications. Dexmedetomidine mainly inhibits the release of norepinephrine by acting on the α-adrenergic receptor of the brainstem nucleus, which can produce good sedative effects. Hydromorphone has a longer duration of action than fentanyl, and it also has a certain sedative effect. The combination of the two is more conducive to the management of postanesthetic agitation and pain. This study was to compare the effect of different doses of dexmedetomidine combined with hydromorphone in the sedation and analgesia after pediatric tonsillectomy and adenoidectomy.

DETAILED DESCRIPTION:
The computer generates random numbers to allocate patients into different group. Trained research staff who are not involved in the study collect the data. The observer who only stayed in PACU was blinded to the allocation and responsible to record the data.

The primary measurement are pain scores, PAED scores, coughing was evaluated on a 9-point scale (1= no coughing, 2= minimal coughing, one or two times, 3-4= moderate coughing, 3-4 times, 5-6= moderate coughing, more than 5 times, 7-8= severe coughing, more than 10 times, 9= laryngospasm), and extubation time. The secondary measurements are the time to discharge from the post-anaesthesia care unit, and the number of postoperative desaturation.

A sample size of 57 was determined by analysis based on the assumption of the decline of extubation time from other similar study and α=0.05,β=0.2.

The continuous variables were presented as means ± SD and the categorical variables were expressed as frequency.

The outcome of interest is extubation time decline.

ELIGIBILITY:
Inclusion Criteria:

* experienced tonsillectomy and adenoidectomy
* ASA physical status I-II
* weight 12-30 kg

Exclusion Criteria:

* respiratory disease
* circulatory or nervous system disease
* hepatic dysfunction
* known adverse reactions to hydromophine and dexmedetomidine

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2019-02-10 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
extubation time | duration from the time that patients arrived in PACU to the time of extubation, though study completion, average 40 mins
  the time of extubation after surgery
Agitation scores | scores at the time point of 0 minute after extubation
  pediatric anesthesia emergence delirium (PAED) scores included five behaviors:(1)makes eye contact with caregiver,(2) actions are purposeful,(3) aware of surroundings,(4) restless,(5) inconsolable.
  Each behavior was correlated to different degree(4= not at all,3= just a little, 2= quite a bit, 1= very much,0= extremely). The scores for each of the five listed behaviors are added to achieve a total score (maximum score of 20, minimum score of 0). A score of >12 is diagnosed to agitation.
Agitation scores | scores at the time point of 5 minutes after extubation
  pediatric anesthesia emergence delirium (PAED) scores included five behaviors:(1)makes eye contact with caregiver,(2) actions are purposeful,(3) aware of surroundings,(4) restless,(5) inconsolable.
  Each behavior was correlated to different degree(4= not at all,3= just a little, 2= quite a bit, 1= very much,0= extremely). The scores for each of the five listed behaviors are added to achieve a total score (maximum score of 20, minimum score of 0). A score of >12 is diagnosed to agitation.
Agitation scores | scores at the time point of 10 minutes after extubation
  pediatric anesthesia emergence delirium (PAED) scores included five behaviors:(1)makes eye contact with caregiver,(2) actions are purposeful,(3) aware of surroundings,(4) restless,(5) inconsolable.
  Each behavior was correlated to different degree(4= not at all,3= just a little, 2= quite a bit, 1= very much,0= extremely). The scores for each of the five listed behaviors are added to achieve a total score (maximum score of 20, minimum score of 0). A score of >12 is diagnosed to agitation.
Agitation scores | scores at the time point of 15 minutes after extubation
  pediatric anesthesia emergence delirium (PAED) scores included five behaviors:(1)makes eye contact with caregiver,(2) actions are purposeful,(3) aware of surroundings,(4) restless,(5) inconsolable.
  Each behavior was correlated to different degree(4= not at all,3= just a little, 2= quite a bit, 1= very much,0= extremely). The scores for each of the five listed behaviors are added to achieve a total score (maximum score of 20, minimum score of 0). A score of >12 is diagnosed to agitation.
coughing score | scores at the time point of 0 minute after extubation
  a 4-point scale that is used to measure severity of coughing(maximum score of 4, minimum score of 1):1= no coughing,2=minimal coughing, one or two times,3= moderate coughing,3-4 times,4= severe coughing, more than 5 times.
coughing score | scores at the time point of 5 minutes after extubation
  a 9-point scale (1= no coughing, 2= minimal coughing, one or two times, 3-4= moderate coughing, 3-4 times, 5-6= moderate coughing, more than 5 times, 7-8= severe coughing, more than 10 times, 9= laryngospasm).
coughing score | scores at the time point of 10 minutes after extubation
  a 9-point scale (1= no coughing, 2= minimal coughing, one or two times, 3-4= moderate coughing, 3-4 times, 5-6= moderate coughing, more than 5 times, 7-8= severe coughing, more than 10 times, 9= laryngospasm).
coughing score | scores at the time point of 15 minutes after extubation
  a 9-point scale (1= no coughing, 2= minimal coughing, one or two times, 3-4= moderate coughing, 3-4 times, 5-6= moderate coughing, more than 5 times, 7-8= severe coughing, more than 10 times, 9= laryngospasm)

CONTACTS AND LOCATIONS:
Overall Officials: e ji Jia, M.D., Principal Investigator — Eye and ENT Hospital of Fudan University
Locations (1):
- Anesthesiology Department of Affiliated Eye and ENT Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olutoye OA, Glover CD, Diefenderfer JW, McGilberry M, Wyatt MM, Larrier DR, Friedman EM, Watcha MF. The effect of intraoperative dexmedetomidine on postoperative analgesia and sedation in pediatric patients undergoing tonsillectomy and adenoidectomy. Anesth Analg. 2010 Aug;111(2):490-5. doi: 10.1213/ANE.0b013e3181e33429. Epub 2010 Jul 7. PMID 20610555
- [Result] Brown KA. What we don't know about childhood obstructive sleep apnoea. Paediatr Anaesth. 2001 Jul;11(4):385-9. doi: 10.1046/j.1460-9592.2001.00719.x. No abstract available. PMID 11442853
- [Result] Patel A, Davidson M, Tran MC, Quraishi H, Schoenberg C, Sant M, Lin A, Sun X. Dexmedetomidine infusion for analgesia and prevention of emergence agitation in children with obstructive sleep apnea syndrome undergoing tonsillectomy and adenoidectomy. Anesth Analg. 2010 Oct;111(4):1004-10. doi: 10.1213/ANE.0b013e3181ee82fa. Epub 2010 Aug 12. PMID 20705788
- [Result] Hauber JA, Davis PJ, Bendel LP, Martyn SV, McCarthy DL, Evans MC, Cladis FP, Cunningham S, Lang RS, Campbell NF, Tuchman JB, Young MC. Dexmedetomidine as a Rapid Bolus for Treatment and Prophylactic Prevention of Emergence Agitation in Anesthetized Children. Anesth Analg. 2015 Nov;121(5):1308-15. doi: 10.1213/ANE.0000000000000931. PMID 26332857
- [Derived] Yi W, Li J, Zhuang Y, Wan L, Li W, Jia J. The effect of two different doses of dexmedetomidine to prevent emergence agitation in children undergoing adenotonsillectomy: a randomized controlled trial. Braz J Anesthesiol. 2022 Jan-Feb;72(1):63-68. doi: 10.1016/j.bjane.2021.08.019. Epub 2021 Oct 8. PMID 34627829